CLINICAL TRIAL: NCT06882031
Title: A Randomized, Open Label, Single-Centre, Single-Dose, 4-Period, 4-Treatment Cross-over Study to Evaluate the Pharmacokinetics of Oral Arsenic Trioxide Solution (SDK001) Under Fasting and Fed Conditions, to Compare to Intravenous Arsenic Trioxide, and to Evaluate Interaction With Calcium Carbonate in Patients With Acute Promyelocytic Leukemia.
Brief Title: Evaluate the Pharmacokinetics of Oral Arsenic Trioxide Solution Under Fasting and Fed Conditions, to Compare Intravenous Arsenic Trioxide, in Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SDK Therapeutics, Inc. (Industry)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SDKARS-101; 173343 (Other Grant/Funding Number: SDK Therapeutics, Inc.)
Record Dates: First submitted 2025-01-23; First posted 2025-03-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-07

CONDITIONS: Acute Promyelocytic Leukemia (APL)
Keywords: APL
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute | interventions — Arsenic Trioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1 (Experimental): In this treatment Arm 1, patients will receive one dose of the following interventions one week apart
  * A: IV Arsenic Trioxide under fasted state
  * B: SDK001 under fasted state
  * C: SDK001 under fed state
  * D: SDK001 with calcium carbonate under fasted state
  Interventions: Drug: Treatment A: Arsenic Trioxide (ATO) Intravenous; Drug: Treatment B: SDK001 (Arsenic Trioxide Oral solution) under faster state; Drug: Treatment C: SDK001 (Arsenic Trioxide Oral solution) under fed state; Drug: Treatment D: SDK001 (Arsenic Trioxide Oral solution) with calcium carbonate
- Sequence 2 (Experimental): In this treatment Arm 2, patients will receive one dose of the following interventions one week apart
  * B: SDK001 under fasted state
  * D: SDK001 with calcium carbonate
  * A: IV Arsenic Trioxide under fasted state
  * C: SDK001 under fed state
  Interventions: Drug: Treatment A: Arsenic Trioxide (ATO) Intravenous; Drug: Treatment B: SDK001 (Arsenic Trioxide Oral solution) under faster state; Drug: Treatment C: SDK001 (Arsenic Trioxide Oral solution) under fed state; Drug: Treatment D: SDK001 (Arsenic Trioxide Oral solution) with calcium carbonate
- Sequence 3 (Experimental): In this treatment Arm 3, patients will receive one dose of the following interventions one week apart
  * C: SDK001 under fed state
  * A: IV Arsenic Trioxide under fasted state
  * D: SDK001 with calcium carbonate
  * B: SDK001 under fasted state
  Interventions: Drug: Treatment A: Arsenic Trioxide (ATO) Intravenous; Drug: Treatment B: SDK001 (Arsenic Trioxide Oral solution) under faster state; Drug: Treatment C: SDK001 (Arsenic Trioxide Oral solution) under fed state; Drug: Treatment D: SDK001 (Arsenic Trioxide Oral solution) with calcium carbonate
- Sequence 4 (Experimental): In this treatment Arm 4, patients will receive one dose of the following interventions one week apart
  * D: SDK001 with calcium carbonate
  * C: SDK001 under fed state
  * B: SDK001 under fasted state
  * A: IV Arsenic Trioxide under fasted state
  Interventions: Drug: Treatment A: Arsenic Trioxide (ATO) Intravenous; Drug: Treatment B: SDK001 (Arsenic Trioxide Oral solution) under faster state; Drug: Treatment C: SDK001 (Arsenic Trioxide Oral solution) under fed state; Drug: Treatment D: SDK001 (Arsenic Trioxide Oral solution) with calcium carbonate

INTERVENTIONS:
Drug: Treatment A: Arsenic Trioxide (ATO) Intravenous — 0.15 mg/kg 2-hour IV infusion of ATO administered under fasted state in single dose
Drug: Treatment B: SDK001 (Arsenic Trioxide Oral solution) under faster state — 0.15 mg/kg SDK001 administered orally under fasted state in single dose
Drug: Treatment C: SDK001 (Arsenic Trioxide Oral solution) under fed state — 0.15 mg/kg SDK001 administered orally under fed state (high fat breakfast) in single dose
Drug: Treatment D: SDK001 (Arsenic Trioxide Oral solution) with calcium carbonate — 0.15 mg/kg SDK001 administered orally with calcium carbonate in tablet form (1g) under fasted state in single dose

SUMMARY:
Randomized, Open-Label Study to evaluate the Pharmacokinetics of Oral Arsenic Trioxide Solution (SDK001) under Fasting and Fed Conditions, to Compare to IV Arsenic Trioxide

ELIGIBILITY:
Inclusion Criteria:

-Diagnosis of APL characterized by the presence of the t(15;17) translocation or promyelocytic leukemia/retinoic acid receptor alpha gene expression

Exclusion Criteria:

* Relapsed or refractory APL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
A Randomized, Open Label, Single-Centre, Single-Dose, 4-Period, 4-Treatment Cross-over Study to Evaluate the Pharmacokinetics of Oral Arsenic Trioxide Solution (SDK001) to Intravenous Arsenic Trioxide | Over 4 weeks in maintenance cycle
  Primary Endpoints
  • AUCinf of AsIII (the pharmacologically active species of ATO) for comparison of SDK001 versus IV ATO

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong-Clinical Trial Centre Phase 1 Centre, Hong Kong, Hong Kong